CLINICAL TRIAL: NCT04170348
Title: Daily Vitamin D for Sickle-cell Respiratory Complications
Acronym: ViDAS-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: FDA Office of Orphan Products Development (U.S. Federal Agency)
Responsible Party: Principal Investigator, Margaret T. Lee, Professor of Pediatrics, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AAAS0396; R01FD006372 (FDA)
Record Dates: First submitted 2019-10-01; First posted 2019-11-20 (Actual); Results first posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Sickle Cell Disease; Anemia, Sickle Cell; Anemia, Hemolytic, Congenital; Respiratory Tract Diseases; Respiration Disorders; Acute Chest Syndrome; Lung Diseases; Asthma; Respiratory Tract Infections; Nutrition Disorders; Deficiency Diseases Vitamin; Vitamin D Deficiency
Keywords: Sickle Cell Disease; Acute Chest Syndrome; Respiratory Complication; Vitamin D Deficiency
MeSH Terms: conditions — Anemia, Sickle Cell; Anemia, Hemolytic, Congenital; Respiratory Tract Diseases; Respiration Disorders; Acute Chest Syndrome; Lung Diseases; Asthma; Respiratory Tract Infections; Nutrition Disorders; Avitaminosis; Vitamin D Deficiency | interventions — Cholecalciferol; Administration, Oral

STUDY DESIGN:
Intervention Model Description: Controlled, double-masked, randomized Phase 2 clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking will be performed by the Research Pharmacy; all other research staff and participants will be blinded to allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Daily oral vitamin D3 (Experimental): Oral vitamin D3, 3,333 IU
  Interventions: Drug: Daily oral vitamin D3, 3,333 IU
- Monthly bolus oral vitamin D3 (Active Comparator): Bolus oral vitamin D3, 100,000 IU
  Interventions: Drug: Monthly oral vitamin D3, 100,000 IU; Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Daily oral vitamin D3, 3,333 IU — Oral vitamin D3, 3,333 IU, will be administered daily.
  Other Names: Cholecalciferol for oral administration
  Arms: Daily oral vitamin D3
Drug: Monthly oral vitamin D3, 100,000 IU — Oral vitamin D3, 100,000 IU, will be administered monthly.
  Other Names: Cholecalciferol for oral administration
  Arms: Monthly bolus oral vitamin D3
Drug: Placebo oral tablet — Participants randomized to receive once monthly oral bolus of vitamin D3, will receive placebo on all other days of the month.
  Arms: Monthly bolus oral vitamin D3

SUMMARY:
This study aims to answer the question whether daily oral vitamin D supplementation can reduce the risk of respiratory or lung complications in children and adolescents with sickle cell disease. Respiratory problems are the leading causes of sickness and of death in sickle cell disease. The investigators hypothesize that daily oral vitamin D3, compared to monthly oral vitamin D, will rapidly increase circulating vitamin D3, and reduce the rate of respiratory complications by 50% or more within the first year of supplementation in children and adolescents with sickle cell disease.

This study is funded by the FDA Office of Orphan Products Development (OOPD).

DETAILED DESCRIPTION:
This is a 2-year controlled, double-blind, randomized Phase 2 clinical trial comparing the efficacy in reducing the rate of respiratory events in sickle-cell disease of daily oral vitamin D3 (3,333 IU/d) with monthly bolus oral vitamin D3, (100,000 IU/mo) as a control. The scientific premise of the clinical trial is that circulating concentrations of vitamin D3, the parent compound, are the principal determinant of the anti-infective and immunomodulatory effects of supplementation.

Eligible participants will be initially screened to determine their blood vitamin D levels. Those with 25-hydroxyvitamin D levels between 5 and 60 ng/mL will be assigned by chance to one of the two arms for 24 months. Participants will be checked every month and will have periodic blood and urine tests to monitor for any side effects of the study treatments. Children above 5 y/o who can cooperate and understand the procedure will have lung function test at baseline and at 24 months. Showing that a monthly dose of vitamin D reduces lung infections, asthma and the acute chest syndrome could help establish this simple, low-cost treatment as a way to decrease sickness and deaths in children and adolescents with sickle-cell disease.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of sickle cell disease (Hb SS, Hb SC, Hb S-Beta-thalassemia)
2. Age 3-20 years old

Exclusion Criteria:

1. Patient unwilling or unable to provide written informed consent (and assent, if applicable)
2. Patient unable or unwilling to comply with requirements of the clinical trial
3. Participation in another clinical trial
4. Current diagnosis of rickets
5. History of hypercalcemia or diagnosis of any medical condition associated with hypercalcemia, including primary hyperparathyroidism, malignancy, sarcoidosis, tuberculosis, granulomatous disease, familial hypocalciuric hypercalcemia
6. Current use of corticosteroids, excluding inhaled steroids
7. Current use of anticonvulsants (phenytoin, phenobarbital, carbamazepine)
8. Therapy with thiazide diuretics or lithium carbonate
9. Known liver or renal disease
10. Patients taking medications for pulmonary complications of sickle cell disease not on a stable dose of medications, as defined by a change in medications or doses within the three months prior to study entry
11. Patients on chronic red blood cell transfusion therapy

Ages: 3 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary M Brittenham, MD, Study Chair — Columbia University; Margaret T Lee, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee MT, Kattan M, Fennoy I, Arpadi SM, Miller RL, Cremers S, McMahon DJ, Nieves JW, Brittenham GM. Randomized phase 2 trial of monthly vitamin D to prevent respiratory complications in children with sickle cell disease. Blood Adv. 2018 May 8;2(9):969-978. doi: 10.1182/bloodadvances.2017013979. PMID 29712666
- [Background] Williams KM, Lee MT, Licursi M, Brittenham GM, Fennoy I. Response to Long-term Vitamin D Therapy for Bone Disease in Children With Sickle Cell Disease. J Pediatr Hematol Oncol. 2018 Aug;40(6):458-461. doi: 10.1097/MPH.0000000000001155. PMID 29668535
- [Background] De A, Anekwe CV, Kattan M, Yao Y, Jin Z, Brittenham GM, Lee MT. Validation of a Questionnaire to Identify Respiratory Tract Infections in Children With Sickle Cell Disease. J Pediatr Hematol Oncol. 2021 Jul 1;43(5):e661-e665. doi: 10.1097/MPH.0000000000002164. PMID 33885042

RESULTS

PARTICIPANT FLOW:
Groups:
- Monthly Bolus Oral Vitamin D3: Bolus oral vitamin D3, 100,000 IU
  Bolus oral vitamin D3, 100,000 IU: Bolus oral vitamin D3, 100,000 IU, will be administered monthly.
  Placebo oral tablet: Participants randomized to receive once monthly oral bolus of vitamin D3, will receive placebo on all other days of the month.
Period: Overall Study
Arm/Group | Daily Oral Vitamin D3 | Monthly Bolus Oral Vitamin D3
Started | 27 | 31
Completed | 22 | 23
Not Completed | 5 | 8
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 1 | 5
Not completed — Non-adherence | 1 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Daily Oral Vitamin D3 | Monthly Bolus Oral Vitamin D3 | Total
Number analyzed (Participants) | 27 | 31 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 25 | 30 | 55
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 16 | 28
  Male | 15 | 15 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 17 | 34
  Not Hispanic or Latino | 9 | 12 | 21
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 17 | 28
  White | 4 | 6 | 10
  More than one race | 8 | 4 | 12
  Unknown or Not Reported | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 27 | 31 | 58

OUTCOME MEASURES:

1. Primary Outcome: Annual Rate of Respiratory Events
Description: Respiratory events will be calculated as the sum of respiratory infection, asthma exacerbation, and acute chest syndrome, as ascertained by use of a validated questionnaire.
Time Frame: Month 12, Month 24
Measure: Mean (Standard Deviation); unit: Respiratory events per year
Arm/Group | Daily Oral Vitamin D3 | Monthly Bolus Oral Vitamin D3
Number analyzed (Participants) | 27 | 31
Respiratory events per year
  Treatment Year 1 | 3.3 (2.1) | 3.3 (2.6)
  Treatment Year 2 | 3.4 (1.7) | 3.2 (2.4)

2. Secondary Outcome: Mean Forced Vital Capacity (FVC % Predicted)
Description: This is to measure the forced vital capacity (FVC; % predicted) at baseline and at month 24.
  Forced Vital Capacity (FVC) is a key measure of lung function that indicates the total volume of air a person can forcefully exhale after taking a deep breath. It is calculated using spirometry, which assesses lung capacity and helps diagnose respiratory conditions. Predicted FVC: The FVC is compared to predicted values based on age, height, and sex to determine if it is within the normal range (80% or more of predicted). Interpretation: A low FVC may indicate obstruction (e.g., asthma or COPD), while a high FVC may suggest restriction in lung function. Baseline Measurement: It is essential to establish a baseline FVC to monitor changes over time and assess the effectiveness of treatments. For accurate interpretation, it is crucial to compare FVC results with other measurements, such as FEV1, to identify the presence of obstructive or restrictive lung disease.
Time Frame: Baseline, Month 24
Population: Due to COVID-19 restrictions, data was only collected/analyzed for 13 out of 27 at baseline and 18 out of 27 at month 24 for DAILY ARM; data was collected/analyzed for 14 out of 31 at baseline and 21 out 31 at month 24 for MONTHLY ARM.
Measure: Mean (Standard Deviation); unit: percent predicted
Arm/Group | Daily Oral Vitamin D3 | Monthly Bolus Oral Vitamin D3
Number analyzed (Participants) | 18 | 21
percent predicted
  Baseline: number analyzed (Participants) | 13 | 14
  Baseline | 86.3 (9.4) | 84.3 (13.2)
  Month 24 | 83.2 (9.9) | 88.7 (11.8)

3. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1)
Description: Forced Expiratory Volume in 1 second (FEV1; % predicted) at baseline and at month 24.
Time Frame: Baseline, Month 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent predicted
Arm/Group | Daily Oral Vitamin D3 | Monthly Bolus Oral Vitamin D3
Number analyzed (Participants) | 18 | 21
percent predicted
  Baseline: number analyzed (Participants) | 13 | 14
  Baseline | 84.6 (9.2) | 84.4 (12.5)
  Month 24 | 85.5 (12.6) | 90.8 (12.9)

4. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1)/Forced Vital Capacity Ratio
Description: Forced Expiratory Volume in 1 second (FEV1; % predicted)/Forced Vital Capacity (FVC) [FEV1/FVC] % predicted at baseline and month 24
Time Frame: Baseline, Month 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Daily Oral Vitamin D3 | Monthly Bolus Oral Vitamin D3
Number analyzed (Participants) | 18 | 21
ratio
  Baseline: number analyzed (Participants) | 13 | 14
  Baseline | 97.9 (6.5) | 100.1 (8.0)
  Month 24 | 97.5 (8.0) | 97.7 (9.8)

5. Secondary Outcome: Forced Expiratory Flow at 25%-75% Vital Capacity (FEF25-75, % Predicted)
Description: Forced Expiratory Flow at 25%-75% vital capacity (FEF25-75) % predicted at baseline and month 24 .
Time Frame: Baseline, Month 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent predicted
Arm/Group | Daily Oral Vitamin D3 | Monthly Bolus Oral Vitamin D3
Number analyzed (Participants) | 18 | 21
percent predicted
  Baseline: number analyzed (Participants) | 13 | 14
  Baseline | 80.9 (22.3) | 86.6 (24.8)
  Month 24 | 81.1 (26.5) | 83.7 (25.0)

6. Secondary Outcome: Ratio of Residual Lung Volume (RV) to Total Lung Capacity (TLC)
Description: Ratio of Residual Lung Volume (RV) to Total Lung Capacity (RV/TLC) at baseline and month 24.
Time Frame: Baseline, Month 24
Population: Due to COVID-19 restrictions, data was only collected/analyzed for 11 out of 27 at baseline and 16 out of 27 at month 24 for DAILY ARM; data was collected/analyzed for 12 out of 31 at baseline and 18 out 31 at month 24 for MONTHLY ARM.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Daily Oral Vitamin D3 | Monthly Bolus Oral Vitamin D3
Number analyzed (Participants) | 16 | 18
ratio
  Baseline: number analyzed (Participants) | 11 | 12
  Baseline | 121.0 (28.2) | 101.2 (28.9)
  Month 24 | 106.9 (34.6) | 109.1 (19.0)

7. Secondary Outcome: Diffusing Capacity of the Lungs for Carbon Monoxide (DLCO)
Description: Diffusing Capacity of the Lungs for Carbon Monoxide (DLCO; % predicted) at baseline and month 24
Time Frame: Baseline, Month 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent predicted
Arm/Group | Daily Oral Vitamin D3 | Monthly Bolus Oral Vitamin D3
Number analyzed (Participants) | 16 | 18
percent predicted
  Baseline: number analyzed (Participants) | 11 | 12
  Baseline | 87.3 (10.3) | 85.3 (15.8)
  Month 24 | 86.5 (12.5) | 90.0 (14.1)

8. Secondary Outcome: Neutrophil Count
Description: Blood Neutrophil Count in percentage at baseline, month 12 and month 24
Time Frame: Baseline, Month 12, Month 24
Population: Data was collected and analyzed only for the following numbers of study participants out of 27 for DAILY ARM and 31 for MONTHLY ARM at each time point due to some study participants did not complete the study.
Measure: Mean (Standard Deviation); unit: Percentage of Neutrophils
Arm/Group | Daily Oral Vitamin D3 | Monthly Bolus Oral Vitamin D3
Number analyzed (Participants) | 27 | 31
Percentage of Neutrophils
  Baseline | 45.8 (13.5) | 43.9 (9.6)
  Month 12: number analyzed (Participants) | 22 | 25
  Month 12 | 47.7 (13.8) | 43.0 (11.0)
  Month 24: number analyzed (Participants) | 22 | 23
  Month 24 | 45.5 (14.8) | 46.8 (12.0)

9. Secondary Outcome: Platelet Count
Description: Blood Platelet Count (Platelets*10^3/ per μL) at baseline, month 12 and month 24
Time Frame: Baseline, Month 12, Month 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Platelets *10^3/ per μL
Arm/Group | Daily Oral Vitamin D3 | Monthly Bolus Oral Vitamin D3
Number analyzed (Participants) | 27 | 31
Platelets *10^3/ per μL
  Baseline | 355.1 (191.1) | 376.2 (242.0)
  Month 12: number analyzed (Participants) | 22 | 25
  Month 12 | 390.0 (125.0) | 387.2 (191.8)
  Month 24: number analyzed (Participants) | 22 | 23
  Month 24 | 398.9 (157.3) | 359.9 (150.1)

10. Secondary Outcome: Serum C-reactive Protein (CRP)
Description: Serum C-reactive protein (CRP; mg/L) at baseline, month 12 and month 24
Time Frame: Baseline, Month 12, Month 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Daily Oral Vitamin D3 | Monthly Bolus Oral Vitamin D3
Number analyzed (Participants) | 27 | 31
mg/L
  Baseline | 2.1 (2.6) | 2.9 (3.7)
  Month 12: number analyzed (Participants) | 22 | 25
  Month 12 | 5.9 (13.7) | 3.6 (5.0)
  Month 24: number analyzed (Participants) | 22 | 23
  Month 24 | 3.0 (2.9) | 4.6 (7.9)

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Daily Oral Vitamin D3 | Monthly Bolus Oral Vitamin D3
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/31
Serious Adverse Events (participants affected / at risk) | 8/27 | 3/31
Other Adverse Events (participants affected / at risk) | 23/27 | 19/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daily Oral Vitamin D3 (N=27) | Monthly Bolus Oral Vitamin D3 (N=31)
Pain syndrome (General disorders) | 8 (9) | 3 (3)
Splenic sequestration (Surgical and medical procedures) | 1 (1) | 0 (0)
Acute chest syndrome (General disorders) | 5 (6) | 0 (0)
Bone infection (Infections and infestations) | 1 (1) | 0 (0)
Clinical sepsis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daily Oral Vitamin D3 (N=27) | Monthly Bolus Oral Vitamin D3 (N=31)
Pain syndrome (General disorders) | 20 (50) | 16 (30)
Upper respiratory infection (Infections and infestations) | 9 (17) | 12 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-29): https://cdn.clinicaltrials.gov/large-docs/48/NCT04170348/Prot_SAP_000.pdf